CLINICAL TRIAL: NCT05145517
Title: FLOWGRAFT - A Post-Market Clinical Follow-up Study in Patients Treated With Vascular Grafts
Brief Title: A Post-Market Clinical Follow-up Study in Patients Treated With Vascular Grafts
Acronym: FLOWGRAFT
Status: Recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: FLOWGRAFT
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Vascular Diseases
Keywords: aortic; aneurysm; dissection; stenosis; PAU; IMH
MeSH Terms: conditions — Vascular Diseases; Aneurysm; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Open repair — Open repair of the aorta and peripheral arteries
  Other Names: Open repair of the aorta and peripheral arteries

SUMMARY:
The FLOWGRAFT post-market clinical follow-up study is undertaken to show the safety and performance of FlowWeave Bioseal, FlowNit Bioseal, FlowLine Bipore and FlowLine Bipore Heparin (combined named as Vascular Grafts) in the treatment of arterial diseases, such as dissection, aneurysm, intramural hematoma (IMH), penetrating aortic ulcer (PAU), contained rupture, stenosis in the aorta or peripheral arteries (lower limbs). This includes the use of FlowWeave Bioseal or FlowNit Bioseal for debranching of the head vessels in an alone standing procedure. Furthermore, it includes the use of the FlowLine Bipore and FlowLine Bipore Heparin Grafts as arterious-venous (AV) shunt.

DETAILED DESCRIPTION:
In this study, patients who receive a Vascular Graft for the treatment of arterial diseases (aneurysm, PAU, IMH, dissection, stenosis) of the aorta or peripheral arteries (lower limbs) or as an AV shunt will be observed. This includes patients in whom the Vascular Grafts are used for debranching or reconstruction of the head vessels. Participating physicians will be asked to provide the observations, that were collected during routine care. Written informed consent, specifically allowing the use of clinical records for this observational study, will be obtained from every patient prior to data collection.

The period of data collection will be approximately 60 + 6 months (depending on the date of the last follow-up visit) from the date of intervention for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years at time of written informed consent
* Patient was selected for treatment with a commercially available Vascular Graft of JOTEC
* Patient satisfies at least one of the following categories:

  * Acute (14 days) / subacute (15 - 90 days) dissection with double lumina in the aorta or peripheral artery / arteries (lower limb)
  * Chronic (>90 days) dissection with double lumina in the aorta or peripheral artery / arteries (lower limb)
  * Aneurysm in the aorta or peripheral artery / arteries (lower limb)
  * IMH in the aorta or peripheral artery / arteries (lower limb)
  * PAU in the aorta or peripheral artery / arteries (lower limb)
  * Contained rupture in the aorta or peripheral artery / arteries (lower limb)
  * Stenosis in the aorta or peripheral artery / arteries (lower limb)
  * Debranching of head vessels
  * AV shunt
* Patient is willing and able to comply with all clinical study procedures and study visits.
* Patient has given written informed consent to participate in the study.

Exclusion Criteria:

* Patient has any other medical, social, or psychological problem that in the opinion of the investigator preclude them from receiving this treatment, procedures, and evaluations pre- and post-procedure.
* Patient is scheduled for reconstruction of the tibial artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with arterial disease who are scheduled to be treated with a Vascular Graft according to the instructions for use and their physician's discretion in accordance with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of in-hospital all-cause mortality

SECONDARY OUTCOMES:
All-cause mortality | 30-day, 6-month,12-month, 24-month, 36-month, 60-month
  Rate of all-cause mortality
Vascular Graft-related adverse event | 30-day, 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with Vascular Graft-related adverse event
Freedom from Vascular Graft -related hemorrhage | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with freedom from Vascular Graft -related hemorrhage
Vascular Graft stenosis > 50% or occlusion | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with Vascular Graft stenosis > 50% or occlusion
Vascular Graft primary patency | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with Vascular Graft primary patency
Vascular Graft secondary patency (after reintervention) | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with Vascular Graft secondary patency (after reintervention)
Pseudoaneurysm at the sutures or in the Vascular Graft | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with pseudoaneurysm at the sutures or in the Vascular Graft
Vascular Graft infection | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with vascular Graft infection
New sepsis | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with new sepsis
New stroke | 6-month,12-month, 24-month, 36-month, 60-month
  Rate of patients with new stroke

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Oberhuber, Prof. Dr., Principal Investigator — University hospital Münster
Locations (1):
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No